CLINICAL TRIAL: NCT06754124
Title: Research Assistant
Brief Title: Investigation of the Effects of Pilates Training in Patients With Drug-Resistant Epilepsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Recep Tayyip Erdogan University Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Derya Çağlar, Research Asistant, Recep Tayyip Erdogan University Training and Research Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2024/10
Record Dates: First submitted 2024-12-04; First posted 2024-12-31 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Epilepsy; Cognitive Dysfunction; Seizures; Quality of Life; Sleep; Depression
Keywords: Epilepsy; Cognitive Dysfunction; Seizures; Quality of Life; Sleep; Depression
MeSH Terms: conditions — Epilepsy; Cognitive Dysfunction; Seizures; Depression | interventions — Control Groups

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (13):
- Pilates Group (Experimental): Pilates training will be given individually for approximately 1 hour, 3 days a week for 8 weeks.
  Interventions: Other: Pilates Group
- Control Group (Active Comparator): Routine medication will be continued for 8 weeks.
  Interventions: Other: Control Group
- Evaluation of seizure frequency (No Intervention): Seizure frequency will be calculated based on the patient's diary in the 2 months prior to the assessment. Patients without a seizure diary will be given one and asked to record their seizures for 2 months.
- Evaluation of core stability (No Intervention): "Core" stability was evaluated with two important dimensions, "core" strength and endurance tests.
- Evaluation of balance (No Intervention): Balance will be assessed separately with static and dynamic balance tests. The Balance Error Scoring System test will be used to assess static balance, and the Four-Step Square Test will be used to assess dynamic balance.
- Evaluation of Functional Exercise Capacity (No Intervention): Functional exercise capacity was evaluated using the 6 Minute Walking Test (6-MWT).
- Evaluation of cognitive function (No Intervention): Cognitive function will be assessed with the Standardized Mini Mental State Examination and the Neuropsychological Test Battery for Cognitive Potentials.
- Evaluation of dual task (No Intervention): Dual task will be evaluated by adding a second task to the Timed Up and Go Test (TUG).
- Evaluation of fatigue (No Intervention): Fatigue will be assessed using the Fatigue Severity Scale (FSS).
- Evaluation of kinesiophobia (No Intervention): Kinesiophobia will be assessed with the Tampa Kinesiophobia Scale (TKS).
- Evaluation of sleep quality (No Intervention): Sleep quality will be assessed by the Pittsburgh Sleep Quality Index (PSQI).
- Evaluation of depression (No Intervention): The Inventory of Neurological Disorders Depression in Epilepsy will be used to assess depression.
- Evaluation of quality of life (No Intervention): Quality of Life In Epilepsy (QOLIE-31) will be used to determine health-related quality of life in epilepsy.

INTERVENTIONS:
Other: Pilates Group — Pilates training will be given individually for approximately 1 hour, 3 days a week for 8 weeks. Before starting the exercise training, all participants will be taught the basic elements of Pilates in 1 session. Pilates training will begin with standing exercises for warming up and centering in the supine position. Training will continue with upper and lower extremity movements. The intensity of the exercises will be increased by using different positions and elastic bands. Stretching exercises and posture exercises will be used during the cool-down period. All exercises will start with 10 repetitions and will be increased to 20 later. Each movement will be shown by the physiotherapist first so that the patients can do the movements correctly. The movements that the patients cannot do will be modified appropriately and applied.
  Arms: Pilates Group
Other: Control Group — No exercise will be allowed for 8 weeks and routine medication will continue.
  Arms: Control Group

SUMMARY:
This study was planned to examine the effects of Pilates training in patients with drug-resistant epilepsy. It was planned to include 40 epilepsy patients in the study. The control group was planned to continue routine drug treatment for 8 weeks. The Pilates group was planned to receive Pilates training 3 days a week for 8 weeks in addition to routine drug treatment. It was aimed to examine the effects of Pilates training performed 3 times a week for 8 weeks on seizure frequency, core stability, balance, functional exercise capacity, cognitive functions, dual task, fatigue, kinesiophobia, sleep quality, depression and quality of life in patients with drug-resistant epilepsy.

DETAILED DESCRIPTION:
This study was planned to investigate the effects of Pilates training, a "core" stability-based exercise method that improves body alignment, postural control, and balance in patients with drug-resistant epilepsy, on seizure frequency, core stability, balance, functional exercise capacity, cognitive functions, dual task, fatigue, kinesiophobia, sleep quality, depression, and quality of life. It was planned to include 40 epilepsy patients in the study. The patients were planned to be randomly divided into two groups as Pilates (n: 20) and control (n: 20). The control group was planned to continue routine drug treatment for 8 weeks. The Pilates group was planned to receive Pilates training 3 days a week for 8 weeks in addition to routine drug treatment. Seizure frequency with the seizure diary; the "core" power with the "sit-ups" and the modified "push-ups" tests; the "core" endurans with the lateral bridge, the trunk flexor endurance, the prone bridge and the modified "Biering-Sorensen" tests; balance with the Balance Error Scoring System (BESS) and the Four-Step Square Test (FSTT); functional exercise capacity with the 6-Minute Walk Test (6-MWT); functional mobility and dual task with the Timed Up and Go Test (TUG); cognitive functions with the BILNOT battery; fatigue with the Fatigue Severity Scale (FSS); kinesiophobia with the Tampa Kinesiophobia Scale; sleep quality with the Pittsburgh Sleep Quality Index (PSQI); depression with the Neurological Disorders Depression Inventory in Epilepsy (NDDI); and health-related quality of life with the Quality of Life in Epilepsy Scale (QOLIE-31) were evaluated before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-65
* Being diagnosed with idiopathic refractory epilepsy by a specialist neurologist
* Not having had status epilepticus for 1 year before the study
* Being able to walk independently
* Not having participated in a regular exercise program
* Having a Standardized Mini Mental Test score greater than 24
* Antiepileptic drug doses being stable during the study

Exclusion Criteria:

* History of any diagnosed neurological or neuropsychiatric disease other than epilepsy
* Presence of any cardiovascular, pulmonary, orthopedic or other medical conditions that would limit participation in the study
* Pregnancy and breastfeeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-11-15 (Actual); Primary Completion 2025-06-20 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Evaluation of Physical Activity Level | 8 week
  Physical activity level will be assessed with the long form of the International Physical Activity Questionnaire (IPAQ).
Evaluation of Seizure Frequency | 8 week
  Seizure frequency will be calculated based on the patient's seizure diary for the 2 months prior to the assessment. Patients without a seizure diary will be given a seizure diary and asked to record their seizures for 2 months.
Evaluation of the Strength of "Core" Muscles | 8 week
  Core muscle strength will be assessed with sit-ups and modified push-ups. The number of times individuals can perform each test for 30 seconds will be recorded. Each measurement will be made twice and the best measurement will be used in statistical analysis.
Evaluation of the Endurance of "Core" Muscles | 8 week
  Static endurance of the core muscles will be assessed using the McGill protocol using the lateral bridge test, the Modified Biering-Sorensen trunk extension test, the trunk flexor endurance test, and the prone bridge test. The time that individuals can maintain the test position will be recorded in seconds using a stopwatch. Each measurement will be made twice and the best measurement will be used in the statistical analysis. The test will be terminated when individuals break the test position or say that they cannot continue the test.
Evaluation of Balance | 8 week
  Balance will be assessed separately with static and dynamic balance tests. The Balance Error Scoring System test will be used to assess static balance, and the Four-Step Square Test will be used to assess dynamic balance.
Evaluation of Functional Exercise Capacity | 8 week
  Functional exercise capacity will be assessed with the 6-Minute Walk Test (6-MWT) in accordance with the American Thoracic Society criteria.
Evaluation of Cognitive Function | 8 week
  Cognitive function will be assessed with the Standardized Mini Mental Test and the Neuropsychological Test Battery for Cognitive Potentials.
Evaluation of Dual Task | 8 week
  Dual task will be evaluated by adding a second task to the Timed Up and Go Test. For the motor task, individuals will be asked to carry an empty tray. For the cognitive task, they will be asked to count backwards from 100 by 7s (mental tracking) and to count words starting with the letter A (verbal fluency). The time will be recorded with a stopwatch. The test will be done twice, one as a trial, and the final measurement will be used in statistical analysis.
Evaluation of Fatigue | 8 week
  Fatigue will be assessed using the Fatigue Severity Scale.
Evaluation of Kinesiophobia | 8 week
  Kinesiophobia will be assessed using the Tampa Kinesiophobia Scale.
Evaluation of Sleep Quality | 8 week
  Sleep quality will be assessed using the Pittsburgh Sleep Quality Index.
Evaluation of Depression | 8 week
  The Inventory of Neurological Disorders Depression in Epilepsy will be used to assess depression.
Evaluation of Quality of Life | 8 week
  The Epilepsy Quality of Life Scale will be used to determine health-related quality of life in epilepsy.

CONTACTS AND LOCATIONS:
Overall Officials: Derya CAGLAR, PhD candidate, Study Director — Recep Tayyip Erdogan University Vocational School of Physical Therapy and Rehabilitation
Locations (1):
- Recep Tayyip Erdogan University Vocational School of Physical Therapy and Rehabilitation, Rize, Güneysu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No